CLINICAL TRIAL: NCT01714206
Title: An Open-Label, 2-Period, Crossover Study to Evaluate the Effects of Multiple Doses of JNJ-28431754 on the Pharmacokinetics of Multiple Doses of Digoxin in Healthy Subjects.
Brief Title: A Study to Assess the Effects of Canagliflozin (JNJ-28431754) on the Pharmacokinetics and Safety of Digoxin in Healthy Volunteers.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CR016465; 28431754DIA1014 (Other: Johnson & Johnson Pharmaceutical Research & Development, L.L.C.)
Record Dates: First submitted 2012-10-23; First posted 2012-10-25 (Estimated); Last update posted 2012-11-19 (Estimated); Status verified 2012-11

CONDITIONS: Healthy
Keywords: Healthy; Canagliflozin (JNJ-28431754); Pharmacokinetics; Digoxin (LANOXIN)
MeSH Terms: interventions — Digoxin; Canagliflozin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment A (Active Comparator): Each volunteer will receive digoxin once daily on Days 1 through 7.
  Interventions: Drug: Digoxin 0.5 mg; Drug: Digoxin 0.25 mg
- Treatment B (Experimental): Each volunteer will receive digoxin once daily on Days 1 through 7 in combination with canagliflozin (JNJ-28431754) once daily on Days 1 through 7.
  Interventions: Drug: Digoxin 0.5 mg; Drug: Digoxin 0.25 mg; Drug: Canagliflozin (JNJ-28431754)

INTERVENTIONS:
Drug: Digoxin 0.5 mg — Two 0.25 mg tablets (0.5 mg total dose) taken orally (by mouth) on Day 1.
  Other Names: Lanoxin
Drug: Digoxin 0.25 mg — One 0.25 mg tablet taken orally on Days 2 through 7.
  Other Names: Lanoxin
Drug: Canagliflozin (JNJ-28431754) — One 300 mg tablet taken orally on Days 1 through 7.
  Other Names: JNJ-28431754
  Arms: Treatment B

SUMMARY:
The purpose of this study is to determine how multiple doses of canagliflozin (JNJ-28431754) affect the pharmacokinetics (ie, how the body affects the drug) of multiple doses of digoxin. The safety and tolerability of canagliflozin will also be assessed in healthy volunteers.

DETAILED DESCRIPTION:
This study will be an open label (all volunteers and study staff know the identity of the assigned treatment), randomized (the treatment is assigned by chance), multiple dose, cross-over study (all volunteers will switch from one treatment to another) to determine how canagliflozin (a drug currently being investigated for the treatment of type 2 diabetes mellitus) affects the pharmacokinetics of digoxin (a drug used to treat various heart conditions). Volunteers will be randomly assigned to 1 of 2 treatment sequence groups: Group AB or Group BA. Volunteers assigned to Group AB will be given Treatment A: digoxin once a day for 7 days. Volunteers assigned to Group BA will be given Treatment B: digoxin and canagliflozin once a day for 7 days. A washout period (when no medication is given) of at least 14 days will follow the first 7-day treatment period. Following the washout period, volunteers will be assigned to the treatment that they did not receive during the first treatment period. This second treatment period will last for 7 days. Each volunteer will participate in the study for approximately 60 days.

ELIGIBILITY:
Inclusion Criteria:

* Volunteers must have a body mass index (BMI = weight in kg/height in m2) between 18 and 30 kg/m2 (inclusive), and body weight not less than 50 kg
* Exclusion Criteria:
* History of, or current active illness, considered to be clinically significant by the Investigator, or any other illness that the Investigator considers should exclude the patient from the study, or that could interfere with the interpretation of the study results

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2009-06; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Plasma concentration of digoxin | Days 5 through 7
  Comparison of plasma concentrations of digoxin following administration of digoxin alone (Treatment A) or in combination with canagliflozin (JNJ-28431754) (Treatment B). This will be used to determine whether there is a pharmacokinetic interaction between digoxin and canagliflozin.
Urine concentration of digoxin | Day 7
  Comparison of the urine concentrations of digoxin following administration of digoxin alone (Treatment A) or in combination with canagliflozin (JNJ-28431754) (Treatment B). This will be used to determine whether there is a pharmacokinetic interaction between canagliflozin and digoxin.

SECONDARY OUTCOMES:
There are no secondary outcome measures

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- [Derived] Devineni D, Manitpisitkul P, Vaccaro N, Bernard A, Skee D, Mamidi RN, Tian H, Weiner S, Stieltjes H, Sha S, Rothenberg P. Effect of canagliflozin, a sodium glucose co-transporter 2 inhibitor, on the pharmacokinetics of oral contraceptives, warfarin, and digoxin in healthy participants. Int J Clin Pharmacol Ther. 2015 Jan;53(1):41-53. doi: 10.5414/CP202157. PMID 25345427